CLINICAL TRIAL: NCT03968653
Title: A Phase 1 Study of Oral Debio 0123 in Combination With Carboplatin in Patients With Advanced Solid Tumors
Brief Title: Study of Oral Debio 0123 in Combination With Carboplatin in Participants With Advanced Solid Tumors
Status: Terminated | Phase: Phase 1 | Type: Interventional
Why Stopped: This trial was concluded for strategic reasons.
Sponsor: Debiopharm International SA (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: Debio 0123-101; 2024-510984-52 (Other: EU CTIS); U1111-1302-8405 (Other: WHO Unique Trial identifier)
Record Dates: First submitted 2019-05-28; First posted 2019-05-30 (Actual); Last update posted 2025-12-05 (Actual); Status verified 2025-11

CONDITIONS: Advanced Solid Tumors
Keywords: WEE1-inhibitor
MeSH Terms: interventions — Carboplatin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Dose Escalation: Group A: Debio 0123 (Experimental): Participants will receive Debio 0123 as monotherapy (Day -3), orally, daily for 3 days during Cycle 1 then in combination with carboplatin intravenous infusion from Cycle 2 onwards.
  Depending on pharmacokinetics (PK) and safety results from previous cohorts, the Debio 0123 dosing regimen may be modified for subsequent cohorts.
  Interventions: Drug: Debio 0123; Drug: Carboplatin
- Dose Escalation: Group B: Debio 0123 (Experimental): Participants will receive Debio 0123, orally, daily, for 6 days during each cycle in combination with carboplatin IV infusion.
  Interventions: Drug: Debio 0123; Drug: Carboplatin
- Dose Expansion: Debio 0123 (Experimental): Participants with platinum-resistant selected solid tumors will receive Debio 0123, orally, daily, depending on the RP2D determined in the previous part, for 3 or 6 days during each cycle in combination with carboplatin IV infusion.
  Interventions: Drug: Debio 0123; Drug: Carboplatin

INTERVENTIONS:
Drug: Debio 0123 — Debio 0123 will be given as an oral capsule for 3 days during each 21-day cycle, except Cycle 1 which is of 24 days.
  Arms: Dose Escalation: Group A: Debio 0123
Drug: Carboplatin — Carboplatin will be given as an IV infusion in combination with Debio 0123 on Day 1 from Cycle 2 onwards in Group A.
  Arms: Dose Escalation: Group A: Debio 0123
Drug: Debio 0123 — Debio 0123 will be given as an oral capsule for 3 or 6 days during each 21-day cycle.
  Arms: Dose Escalation: Group B: Debio 0123; Dose Expansion: Debio 0123
Drug: Carboplatin — Carboplatin will be given as an IV infusion in combination with Debio 0123 on Day 1 from Cycle 1 onwards.
  Arms: Dose Escalation: Group B: Debio 0123; Dose Expansion: Debio 0123

SUMMARY:
This study has two parts: Dose Escalation and Dose Expansion. The primary objective of the study, in the Dose Escalation Part is to determine the recommended phase 2 dose (RP2D) of Debio 0123 when administered in combination with carboplatin in participants with advanced solid tumors that recurred or progressed after prior cisplatin or carboplatin containing therapy and for which no standard therapy of proven benefit is available.

The primary objective of the study, in the Dose Expansion Part is to characterize the safety and tolerability of Debio 0123 when administered in combination with carboplatin at the RP2D determined during the dose escalation part of the study and to evaluate the preliminary antitumor activity of Debio 0123 when administered in combination with carboplatin.

ELIGIBILITY:
Inclusion Criteria:

Dose Escalation:

* Histologically or cytologically confirmed locally advanced or metastatic solid and nonbleeding tumors that had recurred or progressed following standard therapy, has not responded to standard therapy or for which no standard therapy of proven benefit is available
* Able and willing to undergo tumor biopsy
* Prior platinum-based therapy (carboplatin or cisplatin).
* Life expectancy of at least 3 months
* ECOG PS 0-1

Dose Expansion:

* Histologically or cytologically confirmed, recurrent solid tumors of selected types.
* Participants must have progressed after at least 1 prior platinum-based line of therapy for advanced/metastatic disease.
* Participants must be platinum resistant (defined as progression within 6 months of completion of their most recent platinum-based chemotherapy). Prior poly (ADP-ribose) polymerase (PARP) inhibitor therapy is allowed. Platinum-based therapy does not need to be the last treatment prior to study entry.
* Measurable disease per Response Evaluation Criteria in Solid Tumors (RECIST) version 1.1
* Documented progressive or recurrent disease according to RECIST 1.1 since the last anti-cancer therapy and prior to study entry
* Able and willing to undergo tumor biopsy
* ECOG PS 0-1
* Life expectancy of at least 3 months

Exclusion Criteria:

Dose Escalation and Dose Expansion:

* History of other malignancies requiring active treatment in the last 6 months
* Brain tumors and/or symptomatic brain metastases
* Receiving other investigating agents
* Presence of significant cardiovascular disease or other co-morbidities such as symptomatic ascites
* Prior exposure to any WEE1 inhibitor

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 76 (Actual)
Dates: Start 2019-07-30 (Actual); Primary Completion 2025-10-23 (Actual); Study Completion 2025-10-23 (Actual)

PRIMARY OUTCOMES:
Dose Escalation: Recommended Phase 2 Dose (RP2D) of Debio 0123 When Administered in Combination with Carboplatin | 2 Cycles i.e., 45 days (Cycle 1 = 24 days; Cycle 2 onwards = 21 day-cycles)
Dose Expansion: Percentage of Participants with Treatment-Emergent Serious Adverse Events (SAEs) | Up to 46 months
Dose Expansion: Percentage of Participants with Treatment Discontinuations and Treatment Modifications Due to Adverse Events (AEs) and Laboratory Abnormalities | Up to 46 months
Dose Expansion: Overall Response Rate (ORR) | From the start of study treatment until disease progression/recurrence is documented or analysis cut-off, whichever occurs first (up to 46 months)

SECONDARY OUTCOMES:
Dose Escalation: Percentage of Participants with Dose Limiting Toxicities (DLTs) of Debio 0123 When Administered in Combination with Carboplatin | 2 Cycles i.e., 45 days (Cycle 1 = 24 days; Cycle 2 onwards = 21 day-cycles)
Dose Escalation: Percentage of Participants with Treatment-Emergent SAEs | Up to 46 months
Dose Escalation: Percentage of Participants with TEAEs and Laboratory Abnormalities | Up to 46 months
Dose Escalation: Percentage of Participants with Treatment Discontinuations and Treatment Modifications Due to Adverse Events (AEs) and Laboratory Abnormalities | Up to 46 months
Dose Escalation: Number of Participants with Changes in Vital Signs | Day 1 of each cycle (up to 46 months) [Group A: Cycle 1 = 24 days, Cycle 2 onwards and all cycles in Group B = 21-day cycles]
Dose Escalation: Number of Participants with Changes in ECG | Up to 46 months
Number of Participants with Change in Eastern Cooperative Oncology Group Performance Status (ECOG PS) | Day 1 of each cycle (up to 46 months) [Group A: Cycle 1 = 24 days, Cycle 2 onwards and all cycles in Group B = 21-day cycles]
Dose Escalation: Group A: Plasma Concentration of Debio 0123 | Day -3 to predose Day 1; postdose at multiple time points from Day 3 to Day 21 in Cycle 1 (Cycle 1 = 24 days), Day 1 on Cycle 2 (Cycle 2 onwards = 21 day-cycles) and subsequent cycles (Up to 46 months)
  The pharmacokinetics (PK) of Debio 0123 will be evaluated in plasma.
Dose Escalation: Group A: Concentration of Debio 0123 in Urine | Day -3 to Day 21 Cycle 1 (Cycle 1 = 24 days)
  The PK of Debio 0123 will be evaluated in urine.
Dose Escalation: Group A: Area Under the Concentration Curve Over the Time 0 to Infinity (AUC∞) of Free Platinum in Plasma Ultrafiltrate of Carboplatin in Combination | Day 1 to Day 21 Cycle 2 (Cycle 2 onwards = 21 day-cycles) and subsequent cycles (Up to 46 months)
Dose Escalation: Group B: Plasma Concentration of Debio 0123 | Cycle 1 to Cycle 3: Days 1 and 10 (cycle length = 21 days)
  The PK of Debio 0123 will be evaluated in plasma.
Dose Escalation: Group B: Concentration of Free Platinum in Plasma of Carboplatin | Cycle 1 Day 1 (cycle length = 21 days)
Dose Escalation: Correlation Between Plasma Concentration of Debio 0123 and Changes in QT Interval Corrected Using Fridericia's Formula (QTcF) | Up to 46 months
Dose Escalation: Tumor Response | From the start of study treatment until disease progression/recurrence is documented or analysis cut-off, whichever occurs first (Up to 46 months)
Dose Escalation: Progression Free-Survival (PFS) | From the start of study treatment until disease progression or death from any cause, whichever occurs first (Up to 46 months)
Dose Escalation: Overall Survival (OS) | From the start of study treatment until death from any cause (Up to 46 months)
Dose Expansion: Best Overall Response (BOR) | From the start of study treatment until disease progression/recurrence is documented or analysis cut-off, whichever occurs first (Up to 46 months)
Dose Expansion: Disease Control Rate | From the start of study treatment until disease progression/recurrence is documented or analysis cut-off, whichever occurs first (Up to 46 months)
Dose Expansion: Number of Participants with Best Change in Tumor Size | From the start of study treatment until disease progression/recurrence is documented or analysis cut-off, whichever occurs first (Up to 46 months)
Dose Expansion: Duration of Response (DOR) | Up to disease progression (Up to 46 months)
Dose Expansion: Time to Progression (TTP) | Time from treatment initiation until objective tumor progression (Up to 46 months)
Dose Expansion: Plasma Concentration of Debio 0123 | Cycle 1 and Cycle 2: Days 1, 3, 8 and 15 (cycle length = 21 days)

CONTACTS AND LOCATIONS:
Locations (8):
- Netherlands (3):
  - University Medical Center Groningen, Groningen
  - Leiden University Medical Center, Dept. of Clinical Oncology, Leiden
  - Radboud university medical center, Nijmegen
- Spain (5):
  - Hospital Vall Hebrón, Unidad de Investigación en Terapia Molecular (UITM), Barcelona
  - Clinica Universidad de Navarra, Madrid
  - Hospital Universitario Virgen de la Victoria, Málaga
  - Clinica Universidad de Navarra - Pamplona, Pamplona
  - Instituto Valenciano de Oncologia, Valencia

IPD SHARING:
Plan to Share IPD: No